CLINICAL TRIAL: NCT04555031
Title: Evaluation of Surface Refractive Index Shift of Kalifilcon A Lenses Compared to Dailies Total 1, Precision 1 and Biotrue ONEday Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ROC2-20-012
Record Dates: First submitted 2020-09-11; First posted 2020-09-18 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Habitual Soft Contact Lens Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- kalifilcon A lenses (Experimental)
  Interventions: Device: kalifilcon A lenses
- Dailies Total 1 (Active Comparator)
  Interventions: Device: Dalies Total 1
- Precision 1 (Active Comparator)
  Interventions: Device: Precision 1
- Biotrue ONEday (Active Comparator)
  Interventions: Device: Biotrue ONEday

INTERVENTIONS:
Device: kalifilcon A lenses — Participant will wear the lens for each timepoint of 5, 10 and 15 minutes. A new lens will be inserted for each timepoint.
  Arms: kalifilcon A lenses
Device: Dalies Total 1 — Participant will wear the lens for each timepoint of 5, 10 and 15 minutes. A new lens will be inserted for each timepoint.
  Arms: Dailies Total 1
Device: Precision 1 — Participant will wear the lens for each timepoint of 5, 10 and 15 minutes. A new lens will be inserted for each timepoint.
  Arms: Precision 1
Device: Biotrue ONEday — Participant will wear the lens for each timepoint of 5, 10 and 15 minutes. A new lens will be inserted for each timepoint.
  Arms: Biotrue ONEday

SUMMARY:
Approximately 20 habitual soft contact lens wearing participants will be enrolled in this unilateral, randomized, double-masked (participant and investigator masked) repeated measures insertion study. All participants will be seen for a Screening/Dispensing Visit at which informed consent will be obtained and eligibility will be assessed. If participants satisfy all eligibility criteria and none of the exclusion criteria, subjects will insert study lenses in random, successive order according to unique randomization schedules that will be provided to each Investigator.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and have full legal capacity to volunteer.
* Physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* No active ocular disease or allergic conjunctivitis.
* Not using any topical ocular medications.
* Willing and able to follow instructions.
* Signed a statement of informed consent.

Exclusion Criteria:

* Participating in a conflicting study in the opinion of the Investigator.
* Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Schafer, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch and Lomb Site 01, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 10 participants. Each of the 10 participants wore each lens type for 5, 10 and 15 minutes in a randomly assigned fashion.
Groups:
- All Participants: Participants wore each lens type for 5, 10 and 15 minutes in a randomly assigned fashion. All participants completed the study. All 10 participants completed kalifilcon A lens wear, all 10 participants completing Dailies Total 1 wear, all 10 participants completed Precision 1 wear, and all 10 participants completed Biotrue ONEday wear. There were 10 participants total who wore each lens type for 5, 10 and 15 minutes each.
Period: Overall Study
Arm/Group | All Participants
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects wore each lens type for 5, 10 and 15 minutes in a randomly assigned fashion.
Groups:
- All Participants: Participants wore each lens type for 5, 10 and 15 minutes in a randomly assigned fashion. All participants completed the study, therefore each participant wore kalifilcon A lens, Dailies Total 1, Precision 1, and Biotrue ONEday. The only way to show demography for each lens is to show the same information for 10 participants that completed kalifilcon A lens wear, the 10 participants that completed Dailies Total 1 wear, the 10 participants that completed Precision 1 wear, and the 10 participants that completed Biotrue ONEday wear, but there are 10 participants total, not the 40 that the demography table would show if the duplicate information is entered for each lens to which a participant was exposed.
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 10

OUTCOME MEASURES:

1. Primary Outcome: Surface Refractive Index Shifts at 5 Minutes
Description: Refractive index is the ratio of velocity of light in a material divided with velocity of light in vacuum. The eye was measured for surface refractive index on the refractometer. The refractive index of a medium is the ratio of the speed of light in vacuum to the speed of light in the medium. It has no units.
Time Frame: 5 minutes
Population: Participants wore each lens type for 5, 10 and 15 minutes in a randomly assigned fashion. The surface refractive index was measured at each timepoint. All participants completed the study. All 10 participants completed kalifilcon A lens wear, all 10 participants completing Dailies Total 1 wear, all 10 participants completed Precision 1 wear, and all 10 participants completed Biotrue ONEday wear. There were 10 participants total who wore each lens type for 5, 10 and 15 minutes each.
Measure: Mean (Standard Deviation); unit: No units
Arm/Group | Kalifilcon A Lenses | Dailies Total 1 | Precision 1 | Biotrue ONEday
Number analyzed (Participants) | 10 | 10 | 10 | 10
No units | 1.4102 (0.00220) | 1.4251 (0.00274) | 1.4188 (0.00380) | 1.3788 (0.00157)

2. Primary Outcome: Surface Refractive Index Shifts at 10 Minutes
Description: as for outcome 1
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: No units
Arm/Group | Kalifilcon A Lenses | Dailies Total 1 | Precision 1 | Biotrue ONEday
Number analyzed (Participants) | 10 | 10 | 10 | 10
No units | 1.4102 (0.00241) | 1.4267 (0.00113) | 1.4182 (0.00286) | 1.3786 (0.00080)

3. Primary Outcome: Surface Refractive Index Shifts at 15 Minutes
Description: as for outcome 1
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: No units
Arm/Group | Kalifilcon A Lenses | Dailies Total 1 | Precision 1 | Biotrue ONEday
Number analyzed (Participants) | 10 | 10 | 10 | 10
No units | 1.4105 (0.00163) | 1.4238 (0.00213) | 1.4188 (0.00306) | 1.3793 (0.00150)

ADVERSE EVENTS:
Time Frame: 4 days
Groups:
- All Participants: Participants wore each lens type for 5, 10 and 15 minutes in a randomly assigned fashion. All participants completed the study. All 10 participants completed kalifilcon A lens wear, all 10 participants completing Dailies Total 1 wear, all 10 participants completed Precision 1 wear, and all 10 participants completed Biotrue ONEday wear. There were 10 participants total who wore each lens type for 5, 10 and 15 minutes each. There are were 0 adverse events total in the 10 participants, therefore there were 0 AEs while each participant wore kalifilcon A lens, 0 AEs while each participant wore Dailies Total 1, 0 AEs while each participant wore Precision 1, and 0 AEs while each participant wore Biotrue ONEday. The same is true for serious AEs.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT04555031/Prot_SAP_000.pdf